CLINICAL TRIAL: NCT00603486
Title: SuperSTAT Noninvasive Blood Pressure Monitor Evaluation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: GE Healthcare (Industry)
Responsible Party: Laura Haubner, MD, University of South Florida
Other Study IDs: CS 348
Record Dates: First submitted 2008-01-07; First posted 2008-01-29 (Estimated); Last update posted 2008-07-23 (Estimated); Status verified 2008-07

CONDITIONS: Non-Invasive Blood Pressure
Keywords: Non-invasive Blood Pressure (NIBP); GE Dinamap; SuperSTAT

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: GE DINAMAP with SuperSTAT algorithm monitor — Apply cuff on a limb, cuff is inflated and deflated, monitor will displays non-invasive blood pressure values (systolic, diastolic, MAP, and pulse rate)

SUMMARY:
The accuracy and/or performance of the GE DINAMAP noninvasive blood pressure (NIBP) monitors may be improved with modifications in software and/or hardware monitoring techniques and/or accessories. When changes are being made to the GE Monitor, testing can be done to evaluate performance of the investigational devices during and/or after product development.

ELIGIBILITY:
Inclusion criteria

* Signed informed consent
* Ability to single or dual monitor NIBP, ECG, and/or SpO2, whether or not already being monitored for any or all of these parameters.

Exclusion Criteria

* Any subject deemed too unstable, at the clinician's discretion, to participate in the study
* Any subject with a cardiac anomaly that would cause a disparity between aortic pressures and the periphery.
* Any subject who cannot tolerate, in the opinion of the clinician, multiple blood pressure measurements
* Known disease state or medical condition that A) compromises circulation to the extremity (ies), B) compromises musculo-skeletal integrity, or C) otherwise contraindicates use of a NIBP cuff and/or SpO2 sensor on an extremity or ECG patches on skin
* Excessive movement or excitability causing false values or no determinations (SP10 accuracy study only)

Max Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates in the NICU and newborn areas and/or infants.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of one of the GE DINAMAP NIBP Monitor algorithms, SuperSTAT NIBP, in neonatal and/or infant subjects. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Laura Haubner, MD, Principal Investigator — University of South Florida
Locations (1):
- GE Healthcare, Tampa, Florida, United States